CLINICAL TRIAL: NCT05289999
Title: Interest of the Virtual Reality as an Analgesic Support and in the Management the Pre-procedural Anxiety in Rheumatology
Acronym: REAVIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CHM-2021/S07/08
Record Dates: First submitted 2022-03-03; First posted 2022-03-22 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-03

CONDITIONS: Radiculopathy
Keywords: epidural injection; virtual reality; pain management; performance anxiety
MeSH Terms: conditions — Radiculopathy; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using the virtual reality headset for the first injection (Experimental): Performing the first ultrasound-guided epidural injection through the sacrococcygeal hiatus using the virtual reality headset, then the second injection following the usual conditions of care without the device
  Interventions: Device: Virtual reality headset for first injection
- Using the virtual reality headset for the second injection (Experimental): Performing the first ultrasound-guided epidural injection through the sacrococcygeal hiatus following the usual conditions of care, then the second injection using the virtual reality headset
  Interventions: Device: Virtual reality headset for second injection

INTERVENTIONS:
Device: Virtual reality headset for first injection — Performing the first ultrasound-guided epidural injection through the sacrococcygeal hiatus using the virtual reality headset
  Arms: Using the virtual reality headset for the first injection
Device: Virtual reality headset for second injection — Performing the second ultrasound-guided epidural injection through the sacrococcygeal hiatus using the virtual reality headset
  Arms: Using the virtual reality headset for the second injection

SUMMARY:
As a part of the current rheumatological practice skills, epidural injections through the sacrococcygeal hiatus take part in the strategy for managing radicular diseases. This technical act is easily performed in an outpatient context since it is a brief procedure, performed under clinical and ultrasound control, with good tolerance. Nevertheless, epidural injections by the way of the sacrococcygeal hiatus can be responsible of anxiety for the patient and meet the definition of pain induced by treatment. Among the non-pharmacological methods that can be offered to the patient in this context, hypnosis and distraction allow psycho-corporal support acting on certain factors influencing the painful experience of the gesture: duration of the gesture, calm and pleasant environment, etc... That is the context in which the use of virtual reality is of interest. Its use in supporting procedures generating induced pain has already been evaluated in several studies, in particular in the fields of surgery and anaesthesiology. The use of a virtual reality device also seems suitable in the context of epidural injections, but this theoretical and plausible interest remains to be demonstrated. To our knowledge, the literature on the use of a virtual reality headset to support invasive procedures in rheumatology remains poorly developed. The objective of this study is therefore to assess the interest of using a virtual reality headset in the support of pain relief and the management of peri-procedural anxiety when performing epidural injections through the sacrococcygeal hiatus.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 years)
* Hospitalized in a day-hospitalization department at the General Hospital of Le Mans
* For whom a diagnosis of radiculalgia with a duration of less than 6 months is made, for which the imaging is compatible with the symptoms according to the clinician's interpretation
* For whom the indication of at least 2 epidural injections by the way of the sacrococcygeal hiatus is retained
* Having never experienced an epidural injection through the sacrococcygeal hiatus
* Patient able and willing to answer the auto-administered surveys
* Person affiliated or beneficiary of a social security
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research) after oral and written information

Exclusion Criteria:

* Patient with comorbidity of epilepsy
* Patient with a contraindication to performing epidural injections through the sacrococcygeal hiatus
* Patient suffering from blindness and / or deafness
* Patient receiving benzodiazepines and / or other sedative treatment
* Pregnant, breastfeeding or parturient woman
* Person deprived of liberty by judicial or administrative decision
* Person under forced psychiatric care
* Person subject to legal protection
* Person unable to express consent
* Patient who had participated in an interventional study during the last 30 days
* Severely impaired physical and / or mental health which, according to the investigator, may affect the compliance of the study participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of peri-procedural anxiety when performing epidural injections through the sacrococcygeal hiatus | Day 7
  Peri-procedural anxiety was measured with State and Trait Anxiety Index (STAI)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France